CLINICAL TRIAL: NCT07373626
Title: Prospective Study on Physical Activity Trends in Cancer Survivors Treated at the 'MOvement and REhabilitation' (MO.RE) Clinic
Brief Title: Physical Activity Trends in Cancer Survivors Treated at the 'MOvement and REhabilitation' Clinic
Acronym: MOREACTIVE2025
Status: Recruiting | Type: Observational
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2025/0112639
Record Dates: First submitted 2026-01-05; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-11

CONDITIONS: Behavior; Motor Activity
Keywords: Physical Activity; Physical Exercise; Onco-hematological patients
MeSH Terms: conditions — Behavior; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
An active lifestyle after a cancer diagnosis can reduce the side effects of treatment and improve quality of life, mental health, and survival. Recent evidence in the literature confirms its benefits across various types and stages of cancer. However, the majority of cancer patients do not reach the recommended levels of physical activity due to physical, psychological, and logistical barriers. It is essential that healthcare professionals provide motivational support and address individual barriers to physical activity through the active involvement of patients, thus promoting the adoption and maintenance of an active lifestyle. To achieve this, personalization of physical activity programs is crucial. For this reason, the MOvement & REhabilitation clinic was established in 2022, where a dedicated physiotherapist provides personalized consultations and educational support to promote physical activity among cancer patients.

This study aims to evaluate the trend over time in the amount of physical activity among cancer patients attending the "MOvement and REhabilitation" (MO.RE) clinic. The study also seeks to assess patient engagement, the amount of resources used to help patients maintain an active lifestyle, and any barriers to physical activity.

DETAILED DESCRIPTION:
An active lifestyle after a cancer diagnosis can lead to a reduction in many of the most common adverse effects of oncological treatments or to an improvement in certain cancer-related symptoms. The review published in April 2025 by Bai et al. systematically analyzed the results of over 50 systematic reviews and meta-analyses of randomized controlled trials (RCTs), confirming the benefits associated with physical activity, such as a reduction in cancer-related fatigue, improvements in quality of life, mental health, and physical function. Physical activity has also been shown to contribute to reducing cancer-specific mortality. The benefits extend across different types of cancer and various stages of the disease, making physical activity a cornerstone of integrated oncological care. However, the majority of cancer survivors do not achieve the levels of aerobic physical activity (PA) recommended by the World Health Organization, namely ≥150 minutes per week of moderate activity or ≥75 minutes of vigorous activity.

The most common barriers include persistent treatment-related side effects (such as fatigue, pain, neuropathy), lack of time, low motivation, limited access to facilities, and insufficient guidance on physical activity from healthcare professionals. In particular, among cancer survivors living with pain, fear of worsening symptoms, lack of personalized recommendations, and low self-efficacy represent significant obstacles to adopting an active lifestyle. Despite these challenges, several key facilitators promoting regular physical activity have been identified. These include the perception of improved physical and mental health, a sense of control, social support (from peers or professionals), and the availability of adaptable programs.

Therefore, to support patients in recognizing that participation in exercise programs is not only valuable but feasible, interaction with healthcare professionals must include not only a recommendation for physical activity but also the exploration of patient-specific barriers and guidance on how to overcome them. Indeed, studies have suggested that patient advice is more likely to be effective if healthcare professionals are trained in behavioral change strategies and can use these skills to provide personalized motivational support Individual preferences are central in choosing the type of physical activity: many patients prefer low-impact activities such as walking, home exercises, and personalized consultations, highlighting the importance of a flexible and adaptable approach. Actively engaging patients in exercise programs improves behavioral outcomes. Patient engagement, understood as informed and shared participation in care decisions, promotes self-efficacy, intrinsic motivation, and the sustainability of healthy behaviors. The Transtheoretical Model of Change (TTM) by Prochaska and DiClemente represents a useful theoretical tool to guide personalized interventions, adapted to different stages of behavioral change-from intention to action and maintenance. According to the TTM, the patient's readiness to change can be assessed by the healthcare professional, facilitating a personalized approach and support for engagement. Depending on whether the patient is in a stage of pre-contemplation, contemplation, determination, or action, the professional's advice or support will differ.

Finally, the importance of personalization in physical activity programs has been widely emphasized in the literature.

Given the incidence and prevalence of cancer, together with increased survival due to improved oncological care, promoting an active lifestyle is increasingly important to help individuals with a history of cancer regain a good quality of life, return to daily activities, and contribute to the prevention of other diseases (e.g., cardiovascular disease) and recurrence.

Like a medication, physical activity must be dosed in terms of intensity, frequency, duration, and tailored to the individual's needs and preferences, as recommended by the ACSM.

For this reason, in August 2022, the MOvement and REhabilitation (MO.RE.) clinic was opened by the MFR unit with the support of the Lodini Association (SENOnALTRO and Amiche del CO.RE. projects), dedicated to people with a history of cancer, at any stage of the care pathway, with the mission of providing consultations with an experienced physiotherapist to personalize a physical activity program based on the individual's characteristics, needs, and ongoing or completed therapies.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cancer
* Age over 18 years
* Signed informed consent
* Patients for whom a physical exercise program can be proposed

Exclusion Criteria:

* Patients for whom the physiatric assessment identifies a need for individual rehabilitative treatment
* Significant language barrier
* Neuropsychological, psychiatric, or cognitive deficits, or clinical conditions that prevent participation in an independent physical activity program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult cancer survivors (≥18 years) accessing the MO.RE. clinic. Eligible participants have a history of cancer, can provide informed consent, and are suitable for a structured physical activity program. Patients requiring individualized rehabilitation, with significant language barriers, or with neurocognitive, psychiatric, or clinical conditions that prevent safe participation in independent physical activity are excluded.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Weekly aerobic activity | baseline, 3 months, 6 months
  Collection of the minutes of aerobic physical activity performed in the previous 7 days

SECONDARY OUTCOMES:
Overall physical activity level | baseline, 3 months, 6 months
  The overall physical activity level will be calculated using the International Physical Activity Questionnaire (IPAQ-SF), both in categorical form (low activity levels, moderate activity levels, high activity levels) and continuos form (MET minutes per week)
Patient engagement | baseline
  The level of patient engagement will be categorical, with the following stages: pre-contemplation, contemplation, determination, action.
Number of session completed | 3 months, 6 months
  The session completed and the monitoring activities will be expressed as a number per patients
Exercise-related adverse events | Baseline to 6 months
  Number and type of adverse events (e.g., falls, fractures, pain exacerbation requiring medication) assessed and attributed to exercise by study clinician.
Change in Pain Intensity | 3 months, 6 months
  Pain will be measured using the NPRS scale (0-10 Numeric Pain Rating Scale)
Barriers to performing physical activity | 3 months, 6 months
  Barriers to performing physical activity (number of patient)
Perceived barriers to physical activity assessed by patient-reported items | 3 months, 6 months
  Perceived barriers to physical activity will be assessed through patient-reported items collected during clinical consultations. Patients will be asked to report the presence and perceived impact of specific barriers to physical activity, including pain and competing commitments (work-related activities or medical appointments). The assessment will be descriptive and based on patient self-report.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda USL IRCCS di Reggio Emilia - Unit of Physical Medicine and Rehabilitation, Reggio Emilia, Italy

REFERENCES:
- [Background] Ester M, Wagoner CW, Dreger J, Chen G, McDonough MH, McNeely ML, Culos-Reed SN. Effectiveness of a Self-Monitoring App in Supporting Physical Activity Maintenance Among Rural Canadians With Cancer After an Exercise Oncology Program: Cluster Randomized Controlled Trial. JMIR Cancer. 2023 Sep 7;9:e47187. doi: 10.2196/47187. PMID 37676714
- [Background] Clifford BK, Mizrahi D, Sandler CX, Barry BK, Simar D, Wakefield CE, Goldstein D. Barriers and facilitators of exercise experienced by cancer survivors: a mixed methods systematic review. Support Care Cancer. 2018 Mar;26(3):685-700. doi: 10.1007/s00520-017-3964-5. Epub 2017 Nov 28. PMID 29185105
- [Background] Campbell KL, Winters-Stone KM, Wiskemann J, May AM, Schwartz AL, Courneya KS, Zucker DS, Matthews CE, Ligibel JA, Gerber LH, Morris GS, Patel AV, Hue TF, Perna FM, Schmitz KH. Exercise Guidelines for Cancer Survivors: Consensus Statement from International Multidisciplinary Roundtable. Med Sci Sports Exerc. 2019 Nov;51(11):2375-2390. doi: 10.1249/MSS.0000000000002116. PMID 31626055
- [Background] Bai XL, Li Y, Feng ZF, Cao F, Wang DD, Ma J, Yang D, Li DR, Fang Q, Wang Y, Jiang XF, Huang DH, Li XY, Guo JK, Zhao N, Li ZT, Ma QP, Wang L, Wu QJ, Gong TT. Impact of exercise on health outcomes in people with cancer: an umbrella review of systematic reviews and meta-analyses of randomised controlled trials. Br J Sports Med. 2025 Jul 1;59(14):1010-1020. doi: 10.1136/bjsports-2024-109392. PMID 40300838